CLINICAL TRIAL: NCT06381947
Title: Efficacy and Safety of Bempedoic Acid in Association With Anti-PCSK9 and Ezetimibe in Statin-intolerant Patients: a Randomized Crossover Trial
Brief Title: Efficacy and Safety of Bempedoic Acid in Association With Anti-PCSK9 and Ezetimibe in Statin-intolerant Patients
Acronym: BESAFE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Gennaro Galasso, Professor, University of Salerno
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19092023
Record Dates: First submitted 2024-03-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Dyslipidemias; Statin Adverse Reaction; Cardiovascular Diseases; Lipid Metabolism Disorders
Keywords: Dyslipidemias; Statin intolerance; PCSK9 inhibitors; Ezetimibe; Bempedoic acid; Cardiovascular risk control
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases; Lipid Metabolism Disorders | interventions — PCSK9 Inhibitors; 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe; alirocumab; evolocumab

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, phase 4, open-label, multicentre, 2-way crossover trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCSK9 inhibitors plus ezetimibe and bempedoic acid (Experimental): Patients in therapy with PCSK9 inhibitors, bempedoic acid and ezetimibe
  Interventions: Drug: Lipid-lowering therapy combination with PCSK9 inhibitors, bempedoic acid and ezetimibe
- PCSK9 inhibitors plus ezetimibe (Experimental): Patients in therapy with PCSK9 inhibitors and ezetimibe
  Interventions: Drug: Lipid-lowering therapy combination with PCSK9 inhibitors and ezetimibe

INTERVENTIONS:
Drug: Lipid-lowering therapy combination with PCSK9 inhibitors, bempedoic acid and ezetimibe — Evaluation of therapy of bempedoic acid with PCSK9 inhibitors and ezetimibe in reducing LDL-C in statin-intolerant patients.
  Other Names: PCSK9 inhibitors, bempedoic acid, ezetimibe, Praluent, Repatha, Nilemdo, Nustendi, Absorcol
  Arms: PCSK9 inhibitors plus ezetimibe and bempedoic acid
Drug: Lipid-lowering therapy combination with PCSK9 inhibitors and ezetimibe — Evaluation of therapy of PCSK9 inhibitors with ezetimibe in reducing LDL-C in statin-intolerant patients.
  Other Names: PCSK9 inhibitors, ezetimibe, Praluent, Repatha, Absorcol
  Arms: PCSK9 inhibitors plus ezetimibe

SUMMARY:
Statin intolerance occurs in up to 15-20% of treated patients. The combined use of Proprotein Convertase Subtilisin/Kexin type 9 (PCSK9) inhibitors with ezetimibe is commonly performed in these patients, and has been associated with an estimated LDL-C reduction of 65-70%. This drug combination may be insufficient to reach the LDL-C target in high- and very-high-risk patients with statin intolerance, also considering the goals recommended by the current international guidelines. Also, PCSK9 inhibitor dosage escalations frequently fail to achieve the target. Doubling the dosage of alirocumab from 75 mg to 150 mg, when administrated as monotherapy, determines a further reduction of only 3,6% of LDL-C serum level. The full dose of Evolocumab (420 mg every two weeks), was approved only in the setting of homozygous familiar hypercholesterolemia.

Bempedoic acid is an oral, once-daily prodrug, metabolized in the liver to an active inhibitor of ATP-citrate lyase, blocking cholesterol synthesis upstream of 3-hydroxy-3-methylglutaryl-coenzyme A reductase and thereby increasing hepatic expression of the LDL receptor and decreasing circulating LDL-C levels.

The CLEAR (Cholesterol Lowering via Bempedoic acid, an ACL-Inhibiting Regimen) Harmony trial demonstrated that bempedoic acid in addition to maximally tolerated statin therapy did not lead to a higher incidence of adverse events compared to placebo and significantly lowered LDL-C levels. In the CLEAR Serenity study, bempedoic acid showed a safe and effective profile compared with placebo in patients with statin intolerance. In the CLEAR Tranquility, it provided an oral therapeutic option complementary to ezetimibe in patients intolerant to high-dose statins who required additional LDL-C lowering.

The synergistic effect of bempedoic acid plus PCSK9 inhibitors has been investigated by one phase 2 trial (NCT03193047), which showed a statistical superiority of bempedoic acid plus evolocumab strategy versus placebo plus evolocumab in terms of percent change in LDL-C up to 2 months. To date, no randomized phase 3 clinical trial have evaluated the effect of bempedoic acid in association with anti-PCSK9 and ezetimibe in statin-intolerant patients not attaining the recommended LDL-C target.

The investigators hypothesized that the association of bempedoic acid with PCSK9 inhibitors and ezetimibe may be safe and effective in reducing LDL-C in statin-intolerant patients.

DETAILED DESCRIPTION:
This is an investigator-initiated, phase 4, open-label, multicentre, 2-way crossover trial. The study will enlist statin-intolerant patients at high-risk and very high-risk of cardiovascular events, not reaching the LDL-C goal recommended by the 2019 ESC/EAS Guidelines for management of dyslipidaemias based on their individual risk estimate. The patients enrolled have to be intolerant to statin and have not changed their hypolipidemic therapy within 6 weeks prior recruitment.

Eligible participants as per the inclusion criteria will be randomized with 1:1 allocation ratio, without restrictions, into two treatment sequences of 12 weeks, respectively, separated by a washout period of 4 weeks.

Being the inclusion criteria of this study highly selective, the rationale behind the crossover design is the lower sample size needed, and the shorter times to complete the enrolment. Furthermore, since the patients will serve as their own controls, the influence by confounders will be reduced. Being the primary endpoint of this study result of laboratory measurements, the investigators assumed the absence of any carryover effect after the washout period of 4 weeks. Moreover, the investigators assumed the absence of any period effect on the study endpoint.

The phase 1 will start at week 0 (P1-0)and stop at week 12 (P1-12); the phase 2 will start at week 16 (P2-0), after the washout period, and stop at week 28 (P2-12).

The two study treatments will be:

* PCSK9 inhibitors (Evolocumab 140 mg or Alirocumab 75 mg or Alirocumab 150 mg) plus Ezetimibe 10 mg plus Bempedoic acid (Treatment A)
* PCSK9 inhibitors (Evolocumab 140 mg or Alirocumab 75 mg or Alirocumab 150 mg) plus Ezetimibe 10 mg (Treatment B) All patients will be randomly assigned to a Treatment A-Treatment B (AB Group) sequence or to a Treatment B-Treatment A (BA Group) sequence.

The investigators will record laboratory and clinical variables at study visits scheduled for weeks 0, 4, 12, 16, 20, 28. Blood samples will be collected and stored at each visit by the participating centres, and analysed by a central core laboratory (University of Salerno).

At the end of the study, the decision to continue or not treatment with bempedoic acid, as well as any other therapeutic decision, will be left to the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* High- or very-high-risk patients who do not reach the recommended LDL-C target despite lipid-lowering pharmacological therapy for primary or secondary prevention (≤70 mg/dl in high-risk patients, ≤55 mg/dl in very-high-risk patients and ≤40 mg/dl in patients with 2 major cardiovascular events within 2 years)
* Patients treated with PCSK9 inhibitors plus ezetimibe for at least 12 weeks
* Patients with statin intolerance, defined as inability to tolerate at least two statins, one at the lowest starting daily dose and another at any daily dose, either due to objectionable symptoms (real or perceived) or abnormal laboratory analysis, temporally related to statin treatment, reversible upon statin discontinuation, reproducible by rechallenge (restarting medication), and excluding other known factors)
* Age ≥18 years

Exclusion Criteria:

* Fasting blood triglycerides greater than or equal to 500 mg/dL
* Body Mass Index (BMI) greater than or equal to 50 kg/m2
* Severe chronic kidney disease (GFR< 30 ml/min) or glomerular nephropathy
* Recent history (<4 weeks) of clinically significant cardiovascular disease or planning to undergo a major surgical or interventional procedure
* Statin assumption (including low/medium dose and low/medium intensity statins)
* Uncontrolled hypertension
* Uncontrolled hypothyroidism or hyperthyroidism
* Liver disease or dysfunction (Child-Pugh B)
* Gastrointestinal conditions or procedures that could affect drug absorption
* Active malignancy
* Unexplained creatine kinase elevations >3 times the upper limit of normal
* Lipid-modifying therapies prohibited: mipomersen within 6 months of screening, lomitapide, or apheresis within 3 months of screening, inhibitor cholesterol ester transfer protein inhibitors within 2 years of screening (with the exception of evacetrapib, which must have been discontinued ≥3 months prior to screening); and red yeast rice extract and berberine-containing products within 2 weeks of screening
* Participation in other studies
* Unavailable to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean percentage change in LDL-C after 12 weeks of treatment | 0 - 12 weeks
  The primary outcome is the mean percentage change in LDL-C after 12 weeks of treatment

SECONDARY OUTCOMES:
Mean absolute change from baseline to week 12 in low-density lipoprotein cholesterol | 0 - 12 weeks
  Secondary outcome measure
Percentage of patients reaching the recommended LDL-C target | 0 - 28 weeks
  Secondary outcome measure
Changes in plasmatic levels of total cholesterol after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of HDL cholesterol after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of non-HDL cholesterol after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of fasting glucose after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of glycated haemoglobin after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of fasting insulinemia after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of HOMA index after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of hs-CRP after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of lipoprotein(a) after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in plasmatic levels of apolipoprotein B after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Changes in PCSK9 serum levels before starting the treatment and after 12 weeks of treatment | 0 - 12 weeks
  Secondary outcome measure
Number of participants with abnormal uric acid level, abnormal AST/ALT level, ALT or AST >3x ULN, and/or unexplained creatine kinase (CK) >3x ULN | 0 - 28 weeks
  Secondary outcome measure
The number and type of adverse events | 0 - 28 weeks
  Secondary outcome measure
MACE at 12 and 28 weeks | 0 - 28 weeks
  Secondary outcome measure intending as MACE "major adverse cardiovascular events"
Rehospitalization at 12 and 28 weeks | 0 - 28 weeks
  Secondary outcome measure intending as MACE "major adverse cardiovascular events"
Death at 12 and 28 weeks | 0 - 28 weeks
  Secondary outcome measure intending as MACE "major adverse cardiovascular events"

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso R, Cuevas A, Cafferata A. Diagnosis and Management of Statin Intolerance. J Atheroscler Thromb. 2019 Mar 1;26(3):207-215. doi: 10.5551/jat.RV17030. Epub 2019 Jan 19. PMID 30662020
- [Background] Nissen SE, Stroes E, Dent-Acosta RE, Rosenson RS, Lehman SJ, Sattar N, Preiss D, Bruckert E, Ceska R, Lepor N, Ballantyne CM, Gouni-Berthold I, Elliott M, Brennan DM, Wasserman SM, Somaratne R, Scott R, Stein EA; GAUSS-3 Investigators. Efficacy and Tolerability of Evolocumab vs Ezetimibe in Patients With Muscle-Related Statin Intolerance: The GAUSS-3 Randomized Clinical Trial. JAMA. 2016 Apr 19;315(15):1580-90. doi: 10.1001/jama.2016.3608. PMID 27039291
- [Background] Cannon CP, Cariou B, Blom D, McKenney JM, Lorenzato C, Pordy R, Chaudhari U, Colhoun HM; ODYSSEY COMBO II Investigators. Efficacy and safety of alirocumab in high cardiovascular risk patients with inadequately controlled hypercholesterolaemia on maximally tolerated doses of statins: the ODYSSEY COMBO II randomized controlled trial. Eur Heart J. 2015 May 14;36(19):1186-94. doi: 10.1093/eurheartj/ehv028. Epub 2015 Feb 16. PMID 25687353
- [Background] Moriarty PM, Thompson PD, Cannon CP, Guyton JR, Bergeron J, Zieve FJ, Bruckert E, Jacobson TA, Kopecky SL, Baccara-Dinet MT, Du Y, Pordy R, Gipe DA; ODYSSEY ALTERNATIVE Investigators. Efficacy and safety of alirocumab vs ezetimibe in statin-intolerant patients, with a statin rechallenge arm: The ODYSSEY ALTERNATIVE randomized trial. J Clin Lipidol. 2015 Nov-Dec;9(6):758-769. doi: 10.1016/j.jacl.2015.08.006. Epub 2015 Aug 29. PMID 26687696
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Roth EM, McKenney JM. ODYSSEY MONO: effect of alirocumab 75 mg subcutaneously every 2 weeks as monotherapy versus ezetimibe over 24 weeks. Future Cardiol. 2015;11(1):27-37. doi: 10.2217/fca.14.82. PMID 25606700
- [Background] Fala L. Repatha (Evolocumab): Second PCSK9 Inhibitor Approved by the FDA for Patients with Familial Hypercholesterolemia. Am Health Drug Benefits. 2016 Mar;9(Spec Feature):136-9. No abstract available. PMID 27668060
- [Background] Honigberg MC, Natarajan P. Bempedoic Acid for Lowering LDL Cholesterol. JAMA. 2019 Nov 12;322(18):1769-1771. doi: 10.1001/jama.2019.16598. No abstract available. PMID 31714973
- [Background] Ray KK, Bays HE, Catapano AL, Lalwani ND, Bloedon LT, Sterling LR, Robinson PL, Ballantyne CM; CLEAR Harmony Trial. Safety and Efficacy of Bempedoic Acid to Reduce LDL Cholesterol. N Engl J Med. 2019 Mar 14;380(11):1022-1032. doi: 10.1056/NEJMoa1803917. PMID 30865796
- [Background] Laufs U, Banach M, Mancini GBJ, Gaudet D, Bloedon LT, Sterling LR, Kelly S, Stroes ESG. Efficacy and Safety of Bempedoic Acid in Patients With Hypercholesterolemia and Statin Intolerance. J Am Heart Assoc. 2019 Apr 2;8(7):e011662. doi: 10.1161/JAHA.118.011662. PMID 30922146
- [Background] Ballantyne CM, Banach M, Mancini GBJ, Lepor NE, Hanselman JC, Zhao X, Leiter LA. Efficacy and safety of bempedoic acid added to ezetimibe in statin-intolerant patients with hypercholesterolemia: A randomized, placebo-controlled study. Atherosclerosis. 2018 Oct;277:195-203. doi: 10.1016/j.atherosclerosis.2018.06.002. Epub 2018 Jun 12. PMID 29910030
- [Background] Mayne J, Dewpura T, Raymond A, Cousins M, Chaplin A, Lahey KA, Lahaye SA, Mbikay M, Ooi TC, Chretien M. Plasma PCSK9 levels are significantly modified by statins and fibrates in humans. Lipids Health Dis. 2008 Jun 11;7:22. doi: 10.1186/1476-511X-7-22. PMID 18547436
- [Background] Berge KE, Ose L, Leren TP. Missense mutations in the PCSK9 gene are associated with hypocholesterolemia and possibly increased response to statin therapy. Arterioscler Thromb Vasc Biol. 2006 May;26(5):1094-100. doi: 10.1161/01.ATV.0000204337.81286.1c. Epub 2006 Jan 19. PMID 16424354
- [Background] Welder G, Zineh I, Pacanowski MA, Troutt JS, Cao G, Konrad RJ. High-dose atorvastatin causes a rapid sustained increase in human serum PCSK9 and disrupts its correlation with LDL cholesterol. J Lipid Res. 2010 Sep;51(9):2714-21. doi: 10.1194/jlr.M008144. Epub 2010 Jun 5. PMID 20525997
- [Background] Davignon J, Dubuc G. Statins and ezetimibe modulate plasma proprotein convertase subtilisin kexin-9 (PCSK9) levels. Trans Am Clin Climatol Assoc. 2009;120:163-73. PMID 19768174
- [Background] Kastelein JJ, Ginsberg HN, Langslet G, Hovingh GK, Ceska R, Dufour R, Blom D, Civeira F, Krempf M, Lorenzato C, Zhao J, Pordy R, Baccara-Dinet MT, Gipe DA, Geiger MJ, Farnier M. ODYSSEY FH I and FH II: 78 week results with alirocumab treatment in 735 patients with heterozygous familial hypercholesterolaemia. Eur Heart J. 2015 Nov 14;36(43):2996-3003. doi: 10.1093/eurheartj/ehv370. Epub 2015 Sep 1. PMID 26330422
- [Background] Kereiakes DJ, Robinson JG, Cannon CP, Lorenzato C, Pordy R, Chaudhari U, Colhoun HM. Efficacy and safety of the proprotein convertase subtilisin/kexin type 9 inhibitor alirocumab among high cardiovascular risk patients on maximally tolerated statin therapy: The ODYSSEY COMBO I study. Am Heart J. 2015 Jun;169(6):906-915.e13. doi: 10.1016/j.ahj.2015.03.004. Epub 2015 Mar 13. PMID 26027630
- [Background] Bays H, Gaudet D, Weiss R, Ruiz JL, Watts GF, Gouni-Berthold I, Robinson J, Zhao J, Hanotin C, Donahue S. Alirocumab as Add-On to Atorvastatin Versus Other Lipid Treatment Strategies: ODYSSEY OPTIONS I Randomized Trial. J Clin Endocrinol Metab. 2015 Aug;100(8):3140-8. doi: 10.1210/jc.2015-1520. Epub 2015 Jun 1. PMID 26030325
- [Background] Farnier M, Jones P, Severance R, Averna M, Steinhagen-Thiessen E, Colhoun HM, Du Y, Hanotin C, Donahue S. Efficacy and safety of adding alirocumab to rosuvastatin versus adding ezetimibe or doubling the rosuvastatin dose in high cardiovascular-risk patients: The ODYSSEY OPTIONS II randomized trial. Atherosclerosis. 2016 Jan;244:138-46. doi: 10.1016/j.atherosclerosis.2015.11.010. Epub 2015 Nov 14. PMID 26638010
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Bray GA. Medical consequences of obesity. J Clin Endocrinol Metab. 2004 Jun;89(6):2583-9. doi: 10.1210/jc.2004-0535. PMID 15181027
- [Background] Masson W, Lobo M, Lavalle-Cobo A, Masson G, Molinero G. Effect of bempedoic acid on new onset or worsening diabetes: A meta-analysis. Diabetes Res Clin Pract. 2020 Oct;168:108369. doi: 10.1016/j.diabres.2020.108369. Epub 2020 Aug 20. PMID 32827596
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Tripathy D, Almgren P, Tuomi T, Groop L. Contribution of insulin-stimulated glucose uptake and basal hepatic insulin sensitivity to surrogate measures of insulin sensitivity. Diabetes Care. 2004 Sep;27(9):2204-10. doi: 10.2337/diacare.27.9.2204. PMID 15333485
- [Background] Dwan K, Li T, Altman DG, Elbourne D. CONSORT 2010 statement: extension to randomised crossover trials. BMJ. 2019 Jul 31;366:l4378. doi: 10.1136/bmj.l4378. PMID 31366597
- [Result] Fitchett DH, Hegele RA, Verma S. Cardiology patient page. Statin intolerance. Circulation. 2015 Mar 31;131(13):e389-91. doi: 10.1161/CIRCULATIONAHA.114.013189. No abstract available. PMID 25825402
- See also: Related Info — https://clinicaltrials.gov/ct2/show/study/NCT03193047

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT06381947/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT06381947/ICF_001.pdf